CLINICAL TRIAL: NCT04547530
Title: A Randomized Double-blind Placebo-controlled Trial to Investigate the Effect of Vitamin D Supplementation in Live Birth Rate of in Vitro Fertilization Outcome
Brief Title: Effect of Vitamin D Supplementation in Live Birth Rate of in Vitro Fertilization Outcome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Kwong Wah Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW19-411
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Active Comparator): Vitamin D 50,000IU per week for 4 weeks from recruitment, followed by 50,000IU per week every 2 weeks throughout the IVF cycle. Subjects to stop own supplements and folic acid will be provided. If pregnant and fetal viability confirmed at 6 weeks gestation, switch to Materna until delivery.
  If not pregnant, to continue vitamin D 50,000IU once every 2 weeks until 6 months from recruitment.
  The rest of the IVF, embryo transfer procedure and antenatal care will be the same as usual practice.
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Placebo tablets identical to the active drug for 4 weeks from recruitment, followed by placebo tablets once every 2 weeks throughout the IVF cycle. Subjects to stop own supplements and folic acid will be provided. If pregnant and fetal viability confirmed at 6 weeks gestation, switch to Materna until delivery.
  If not pregnant, to continue placebo tablets once every 2 weeks until 6 months from recruitment.
  The rest of the IVF, embryo transfer procedure and antenatal care will be the same as usual practice.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — as above
  Arms: Vitamin D
Dietary Supplement: Placebo — as above
  Arms: Placebo

SUMMARY:
This is a randomized-controlled trial evaluating the effect of the use of vitamin D supplementation on the live birth rate in women undergoing in vitro fertilization (IVF). The hypothesis is that administration of vitamin D can increase the live birth rate for women undergoing IVF.

DETAILED DESCRIPTION:
Patients undergoing IVF treatment cycle at Queen Mary Hospital and Kwong Wah Hospital will be invited to participate in this study. Participating subjects will be randomized into either (i) vitamin D or (ii) placebo group in a 1:1 allocation ratio by computer-generated random numbers one month before IVF.

Subjects allocated to the vitamin D group will take vitamin D 50,000IU per week from recruitment for 4 weeks, followed by 50,000IU once every 2 weeks throughout the IVF cycle until fetal viability is confirmed at 6 weeks (if pregnant), after which they will be switched to Materna. If not pregnant, they will continue Vitamin D 50,000IU once every 2 weeks until 6 months from randomization, during which they can undergo frozen-thawed embryo transfer.

Subjects allocated to the placebo group will take placebo tablets which will be identical to the active drug. If pregnant and fetal viability is confirmed at 6 weeks, they will be switched to Materna. If not pregnant, they will continue the placebo tablets until 6 months from randomization, during which they can undergo frozen-thawed embryo transfer.

The clinician and patients will both be blinded to the randomization throughout the course of treatment. The live birth rate of the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women undergoing IVF
* Aged between 18 and 43 years old, inclusive, at the time of signing informed consent
* Having given voluntary written informed consent

Exclusion Criteria:

* Already taking vitamin D
* Undergoing preimplantation genetic testing
* Use of donor oocytes or donor embryos
* Presence of hydrosalpinx not corrected surgically
* Active tuberculosis/ receiving therapy for tuberculosis
* History of any medical condition or medications that may predispose to vitamin D sensitivity, altered vitamin D metabolism and/or hypercalcemia, including history of renal/ureteral stones, parathyroid disease, renal or liver failure, current use of anticonvulsants, current use of steroid
* Allergy to vitamin D
* Abnormal serum calcium values

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1150 (Estimated)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 10 months
  per embryo transfer procedure

SECONDARY OUTCOMES:
Cumulative pregnancy rate within 6 months of randomization | 6 months
  within 6 months of randomization
Serum and follicular vitamin D levels | 6 weeks
  vitamin D levels
Pregnancy rate | 8 weeks
  pregnancy test positive
Clinical pregnancy rate | 10 weeks
  Presence of intrauterine gestational sac on ultrasound
Ongoing pregnancy rate | 12 weeks
  Viable pregnancy beyond 8 weeks
Adverse events | 6 months
  Number of women with adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Kwong Wah Hospital, Hong Kong
  - Queen Mary Hospital, University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided